CLINICAL TRIAL: NCT03210415
Title: Study on Prevention, Treatment and Mechanism of Preterm Labor for Chinese Pregnant Women ≥35 Years Old
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hongbo Qi, Principle Investigator, Ministry of Science and Technology of the People´s Republic of China
Other Study IDs: 2016YFC1000407
Record Dates: First submitted 2017-05-04; First posted 2017-07-07 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Preterm Labor
Keywords: Preterm Labor; China; Pregnant Women; ≥35 Years Old
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, hair, cervical secretion，saliva，amniotic fluid, placenta
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Pregnant women ≥35 years old would have spontaneous preterm labor. There's no intervention in this group, because it's an Observational Study Model.
  Interventions: Other: Observational Study Model
- Control group: Pregnant women ≥35 years old would not have spontaneous preterm labor. There's no intervention in this group, because it's an Observational Study Model.
  Interventions: Other: Observational Study Model

INTERVENTIONS:
Other: Observational Study Model — There is no intervention for the study.

SUMMARY:
In China, there's no effective prevention and treatment on preterm birth for pregnant women ≥35 years old, so this study is necessary.

DETAILED DESCRIPTION:
Because the policy of "Two-child" in China, there are more and more women more than 35 years old choose to have another baby. It is necessary to find out a way to prevent them who is older than 35 from preterm labor. About 1500 pregnant women will be recruited at about gestational age of 14 weeks for this study. All of them will be taken samples (i.e. blood, hair, cervical secretion ) to be saved before and after delivery. After all data collected, the investigators will do analysis of all data and find out strategy and mechanism of preterm labor.

ELIGIBILITY:
Inclusion Criteria:

* Chinese pregnant women ≥ 35 years old

Exclusion Criteria:

* twins or multiple pregnancies, indicated preterm birth, <35 years old, gestational ages ≥ 37 weeks, incomplete data of prenatal care。

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — study on pregnant women
Study Population: Chinese pregnant women ≥ 35 years old with spontaneous preterm birth between 28-37 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity of Preterm birth | 1 years
  Preterm delivery (PTD) is one of the most common and most serious complications of pregnancy. In China, preterm delivery is defined as delivery after 28 weeks completed but before 37 weeks of gestation. PTD rate varies between 5-18 %. Outcome also varies with the quality of neonatal care. create the highest burden for the society.

SECONDARY OUTCOMES:
Social Burden | 1 years
  Outcome varies with the quality of neonatal care. create the highest burden for the society. A 2006 report from the Institute of Medicine estimated the annual cost of preterm birth in the United States to be $26.2 billion or more than $51,000 per premature infant .
Morbidity of Chorioamnionitis | 1 years
  The main hypothesis of the etiology of spontaneous PTD is ascending infection from the lower genital tract up in the sterile uterus invading the decidua, chorioamniotic membranes, amniotic fluid and, in some cases, the fetus. This is responsible for an inflammatory condition that might trigger myometrial contractions, rupture of the membranes and cervical maturation leading to PTD. Investigations have shown that the amount of bacteria present in the amniotic fluid is correlated to the level of intrauterine inflammation. Inflammation is also related to the presence of bacteria in the amniotic fluid and to histological chorioamnionitis.
Respiratory distress syndrome, ischemic hypoxic encephalopathy, necrotizing enterocolitis, various infections | 1 years
  the short-term outcomes of the preterm delivery, which will cost money, time and source to beat. The treatment is not satisfactory, but create the highest burden for the society.
Cerebral palsy, chronic lung disease, blindness caused by retinopathy, auditory nerve abnormalities, mental retardation | 1 years
  the long-term outcomes of the preterm delivery. The main areas that are affected are the respiratory function and the neurodevelopment of these babies due to the early arrest in the lung and brain development, respectively. Moreover, the overall general health of this population is affected in the long-term and ongoing follow up studies are required to provide a better understanding in the field.

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo bo Qi, Dr., Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affilliated Hospital of Chongqig Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464